CLINICAL TRIAL: NCT02464865
Title: Thiamin Deficiency in Obese Thai Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Si656/2014
Record Dates: First submitted 2015-05-18; First posted 2015-06-08 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Obesity; Child; Thiamine Deficiency
Keywords: thiamine deficiency; obese children; Thai
MeSH Terms: conditions — Obesity; Thiamine Deficiency | interventions — Thiamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Thiamine 1 (Experimental): presence of severe symptoms and signs of thiamine deficiency: heart failure, convulsion, coma, loss of ankle and knee jerks with muscular wasting and paralysis (typically symmetrical foot- and wrist-drop)
  Interventions: Drug: Thiamine 1
- Non-thiamine (Other): no symptoms and signs of thiamine deficiency
  Interventions: Other: Non-thiamine
- Thiamine 2 (Experimental): presence of mild symptoms and signs of thiamine deficiency; peripheral neuropathy alone (paraesthesia of hands and feet)
  Interventions: Drug: Thiamine 2

INTERVENTIONS:
Drug: Thiamine 1 — If severe symptoms and signs of thiamine deficiency are present, thiamine is prescribed.
  Intervention 1 : severe symptom (heart failure, convulsion, or coma) : 50 mg thiamin administered very slowly intravenously, followed by a daily intramuscular dose of 10 mg for a week, and finally followed by 3-5 mg of thiamine per day orally for at least 6 weeks
  Arms: Thiamine 1
Other: Non-thiamine — no symptoms and signs of thiamine deficiency
  Arms: Non-thiamine
Drug: Thiamine 2 — If symptoms and signs of thiamine deficiency are present, thiamine is prescribed.
  If mild symptom : a daily oral dose of 10 mg thiamin during the first week, followed by 3-5 mg of thiamin per day orally for at least 6 weeks
  Arms: Thiamine 2

SUMMARY:
This study is aimed to assess the prevalence of thiamin deficiency in obese Thai children.

DETAILED DESCRIPTION:
This study is a cross-sectional study. The objectives of the study are to determine the prevalence of thiamin deficiency in obese Thai children and to assess the associations of dietary factors and thiamin deficiency.

ELIGIBILITY:
Inclusion Criteria:

* obese : weight for height > median + 3 standard deviations
* simple obesity

Exclusion Criteria:

* pathological obesity
* chronic diseases e.g. cerebral palsy, metabolic disease, etc.
* diseases of red blood cells
* on medication e.g. steroid, multivitamins, thiamine-containing vitamins, diuretic drugs
* hemodialysis or peritoneal dialysis
* bariatric surgery

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 124 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
abnormal thiamin pyrophosphate effect | 7 days
  Thiamin pyrophosphate effect will be measured by a blood test

SECONDARY OUTCOMES:
consumption of thiaminase-containing foods and thiamin antagonist-containing foods | 7 days
  Food diary and food frequency questionaire will be required to evaluate food consumption

CONTACTS AND LOCATIONS:
Overall Officials: Narumon Densupsoontorn, MD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkok, Thailand

REFERENCES:
- [Result] Densupsoontorn N, Jirapinyo P, Kangwanpornsiri C. Micronutrient deficiencies in obese Thai children. Asia Pac J Clin Nutr. 2013;22(3):497-503. doi: 10.6133/apjcn.2013.22.3.06. PMID 23945419